CLINICAL TRIAL: NCT02759822
Title: Haploidentical Hematopoietic Stem Cell Transplantation for Acute Leukemias
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Leonardo Javier Arcuri (Other Government)
Responsible Party: Sponsor-Investigator, Leonardo Javier Arcuri, Physician, Instituto Nacional de Cancer, Brazil
Organization: Instituto Nacional de Cancer, Brazil (Other Government)
Other Study IDs: CEMO/INCA-Haplo-01
Record Dates: First submitted 2016-04-22; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma
Keywords: Haploidentical Hematopoietic Stem Cell Transplantation; Partially Matched Hematopoietic Stem Cell Transplantation; Post-transplant Cyclophosphamide; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Acute Lymphoblastic Leukemia: Haploidentical Stem Cell Transplantation with Post Transplant Cyclophosphamide (PTCy)
  Preferred conditioning:
  * Total Body Irradiation 1200 cGy (TBI1200) + Fludarabine 120 mg/m2 (Flu120)
  Alternative conditionings:
  1. Melphalan 100-140 mg/m2 (Mel100-140) + Fludarabine 160 mg/m2 (Flu160) + Total Body Irradiation 200 cGy (TBI200)
  2. Busulfan 9.6 mg/kg (Bu9.6) + Fludarabine 150 mg/m2 (Flu150) + TBI200 Graft versus host disease Prophylaxis: Post-Transplant Cyclophosphamide (PTCy) + Tacrolimus (FK) or Cyclosporin (CSA) + Mycophenolate Mofetil (MMF)
  Interventions: Procedure: Haploidentical Stem Cell Transplantation
- Group B: Acute Myeloid Leukemia: Haploidentical Stem Cell Transplantation with Post Transplant Cyclophosphamide (PTCy) Preferred Conditioning: Mel100-140 + Flu160 + TBI200
  Alternative conditionings:
  1. Bu9,6 + Flu150 + TBI200
  2. Cyclophosphamide 29 mg/kg + Flu150 + TBI200 Graft versus host disease Prophylaxis: PTCy + FK or CSA + MMF
  Interventions: Procedure: Haploidentical Stem Cell Transplantation

INTERVENTIONS:
Procedure: Haploidentical Stem Cell Transplantation — Haploidentical Stem Cell Transplantation from a related donor (partially matched sibling, father, mother, son or daughter).

SUMMARY:
This is a prospective observational cohort study of haploidentical transplantation with post-transplant cyclophosphamide for acute leukemias using reduced intensity conditioning for acute myeloid leukemia (AML) and myeloablative conditioning for acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) is the most effective treatment for acute myeloid leukemia (AML) and acute lymphoblastic leukemia (ALL), with the lowest rates of relapse.

Fertility rate in Brazil is falling, and only 25% of people born today will have a matched sibling donor. On the other hand, currently donor non-related to about 50% of patients enrolled in Brazilian Receptor Registry (REREME). Consequently, at least 35% of patients won't have a matched donor.

The haploidentical transplantation is defined as a partially matched hematopoietic cell transplantation, using a partially matched family donor (parent, sibling or child). Haploidentical transplantation activity is growing worldwide, with results comparable matched unrelated donors.

The objective of this study is to test the feasibility of haploidentical transplantation with post transplant cyclophosphamide for acute leukemias in a Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia or acute myeloid leukemia

Exclusion Criteria:

* Severe comorbidities
* Second transplant

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with acute leukemias referred for stem cell transplantation without HLA-matched related or unrelated donor
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 1 year
  1-year overall survival. Survival curves will be estimated by Kaplan-Meier methodology.

SECONDARY OUTCOMES:
Cumulative incidence of leukemia relapse | 5 years
  Relapse will be defined by reappearance of Leukemic Cells in bone marrow (>5%) or peripheral blood (>1%). Risk factors for leukemia relapse will be estimated by extended Cox Model for competing risks (Fine & Gray model). Competing event will be defined as death in remission.
Transplant Related Mortality | 6 months
  Transplant-related mortality (TRM) will be defined as death in remission. Risk factors for TRM will be estimated by extended Cox Model for competing risks (Fine & Gray model). Competing event will be defined as leukemia relapse.
Cumulative Incidence of acute Graft Versus Host Disease | 5 years
  Acute graft versus host disease will be diagnosed and graded by modified Glucksberg criteria. Risk factor for acute graft versus host disease will be estimated by extended Cox Model for competing risks (Fine & Gray model). Cumulative incidence curves will be estimated by Gray methodology.
Cumulative Incidence of chronic Graft Versus Host Disease | 5 years
  Chronic graft versus host disease will be diagnosed and graded by National Institute of Health Consensus (NIH Consensus). Risk factor for chronic graft versus host disease will be estimated by extended Cox Model for competing risks (Fine & Gray model). Cumulative incidence curves will be estimated by Gray methodology.
Cumulative Incidence of Infectious Complications | 1 year
  Cumulative incidence of viral, fungal and bacterial infections. Subgroups will be compared by Cox Model for competing risks (Fine & Gray model). Cytomegalovirus reactivation will be analyzed by multiple events Cox Model.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo J Arcuri, MD, Principal Investigator — Instituto Nacional de Cancer
Locations (1):
- Instituto Nacional de Cancer, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No